CLINICAL TRIAL: NCT03130465
Title: Aripiprazole Once-monthly Versus Daily Oral Atypical Antipsychotic Treatment in Patients With Recent-onset Schizophrenia: an Observational, Non-interventional Study
Brief Title: Aripiprazole Once-monthly Versus Daily Oral Atypical Antipsychotic Treatment in Patients With Recent-onset Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-303-00136
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: adherence; long-acting injectable antipsychotic; all-cause treatment discontinuation; recent-onset schizophrenia; daily oral atypical antipsychotic
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aripiprazole Once Monthly (AOM): Schizophrenia patients who initiated maintenance treatment with AOM during a schizophrenia-related hospitalisation or during the first three months after this hospitalisation.
- Daily oral atypical AP: Schizophrenia patients who initiated maintenance treatment with any daily oral atypical AP during a schizophrenia-related hospitalisation or during the first three months after this hospitalisation.

SUMMARY:
This is an observational, non-interventional study that will include two cohorts of patients with schizophrenia who initiated maintenance treatment during a schizophrenia-related hospitalisation or during the immediate three months after hospital discharge: patients who initiated maintenance treatment with AOM and patients who initiated maintenance treatment with any daily oral atypical AP.

DETAILED DESCRIPTION:
This is an observational, non-interventional study that will include two cohorts of patients with schizophrenia who initiated maintenance treatment during a schizophrenia-related hospitalisation or during the immediate three months after hospital discharge: patients who initiated maintenance treatment with AOM and patients who initiated maintenance treatment with any daily oral atypical AP.

The date of maintenance treatment initiation will be considered the index date (see definition of maintenance treatment initiation in Section 3.1). Baseline data will be collected immediately after the inclusion of the patient in the study (including retrospective data from the index date to the date of informed consent and from the past 5 years). From the index date, each patient will be followed up until discontinuation of the maintenance treatment of interest and up to a maximum of 12 months. Especially after the implementation of the Global Amendment nº1, it is possible that the complete follow-up of the patient took place in the past (retrospective data), i.e. before the inclusion of the subject in the study. Data will be collected from the patient file and from information obtained during routine visits scheduled according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between ≥18 and ≤35 years of age
2. Diagnosis of schizophrenia confirmed by the current investigator.
3. Initiation of maintenance treatment with AOM (at least one injection) or with daily oral atypical AP before the study start at the site and up to a maximum of 6 months after the launch of AOM in the country, during an inpatient stay due to an acute schizophrenia episode or during the immediate three months after hospital discharge, and prescribed in the usual manner in accordance with the terms of the marketing authorisation.*

   Patients treated in the daycare hospital will be considered:
   * Eligible to be included, if the patient was admitted in the hospital (full time inpatient stay) for an acute psychotic episode and then discharged to a day care hospital in order to achieve stabilization and initiate maintenance antipsychotic treatment. The initiation of the maintenance antipsychotic treatment (index date) must occur before discharge from day care hospital or during the immediate following three months after discharge.
   * NOT eligible, if the patient was treated exclusively in the day care hospital since the first day (i.e. not spending any night at all in the hospital) as these patients are very likely to be subacutely psychotic.

     * The date of initiation of maintenance therapy will be considered the index date. For AOM, it is the date of the first injection. For the oral AP, this date is defined by the physician when patients are believed to be stable enough to be considered "in maintenance treatment".
4. Willingness to participate in the study; subjects must give their written consent to participate unless: they have discontinued treatment or have finished the 12 months follow up period before study inclusion (retrospective assessment only) and a) written consent not required by local regulations, or b) it would take a non-reasonable effort† or c) the source patient is deceased or untraceable.

   * A reasonable effort is defined as 3 contact attempts separated by 3 weeks. All efforts to obtain the informed consent, reasonable or not, shall be registered in the medical history of the patient to be used as documental source.

If allowable by local regulations/Ethics Committees, provision of oral (e.g., by phone) instead of written consent is also possible for patients with retrospective assessment only.

Exclusion Criteria:

1. The patient has a psychiatric disorder other than schizophrenia which is established as the primary diagnosis
2. Chronically hospitalized patients (defined as more than 3 months).
3. Participation in an interventional clinical trial since AOM or daily oral atypical AP were initiated as maintenance treatment or within the previous 6 months to this initiation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible patients will include adult patients (≥18 years) with recent-onset (≤35 years old) schizophrenia who initiated maintenance treatment with AOM or an oral atypical AP during an inpatient stay due to an acute schizophrenia episode or during the immediate three months after hospital discharge and which treatment was initiated before the study start at the site and up to a maximum of 6 months after the launch of AOM in the country. Prescription of the maintenance treatment had to be done in the usual manner in accordance with the terms of the marketing authorisation.
Sampling Method: Probability Sample
Enrollment: 636 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Time (days) to all-cause treatment discontinuation for AOM or daily oral atypical AP | First 12 months after initiation of maintenance treatment
  Treatment discontinuation is defined as the interruption, replacement or addition of a new antipsychotic drug to the main antipsychotic initiated at index date (AOM or daily oral atypical AP).

SECONDARY OUTCOMES:
Treatment discontinuation rate (%) and description of the reasons for treatment discontinuation | First 12 months after initiation of maintenance treatment
  To compare the treatment discontinuation rate and the reasons for this discontinuation during the first 12 months after initiation of maintenance treatment between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP.
Relapse rate (%) in the first 12 months after initiation of maintenance treatment | First 12 months after initiation of maintenance treatment
  To compare the relapse rate in the first 12 months after initiation of maintenance treatment between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP.
Change over time in CGI-S (score) | From index date up to a maximun of 12 months
  To compare the evolution in disease severity according to Clinical Global Impression-Disease Severity (CGI-S) scale from initiation of maintenance treatment and up to the end of follow-up (12 months or up to discontinuation) between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP as maintenance treatment.
Change over time in QLS-5 (score) | From index date up to a maximun of 12 months
  To compare the clinical and functional outcomes according to the 5-item Quality of Life Scale for schizophrenia (QLS-5) from initiation of maintenance treatment and up to the end of follow-up (12 months or up to discontinuation) between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP as maintenance treatment.
All-cause hospitalisation rate (%) in the first 12 months after initiation of maintenance treatment, time to first all-cause hospitalisation and length of hospitalisation(admission/discharge dates) | From index date up to a maximun of 12 months
  To compare all cause hospitalisations in the first 12 months after initiation of maintenance treatment between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP.
Mental health-related hospitalisation rate (%) in the first 12 months after initiation of maintenance treatment, time to first mental health-related hospitalisation and length of mental-health related hospitalisation (admission/discharge dates) | From index date up to a maximun of 12 months
  To compare mental health-related hospitalisations in the first 12 months after initiation of maintenance treatment between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP.
Description of health resource use (HRU) related to schizophrenia (hospitalisations, medications, non-pharmacological therapies, outpatient visits, procedures) | From index date up to a maximun of 12 months
  To compare the health resource use related to schizophrenia in the first 12 months after initiation of maintenance treatment between patients with recent-onset schizophrenia treated with AOM or with a daily oral atypical AP.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (67):
- France (16):
  - H. Paul-Guiraud Clamart, Clamart
  - CH Jonzac, Jonzac
  - Centre Psychotherapique Nancy, Laxou
  - Centre Hospitalier Esquirol, Limoges
  - CHS-La Colombière, Montpellier
  - CHU Nantes Hospital Saint Jacques, Nantes
  - CH Sainte Marie, Nice
  - CHU Pasteur, Nice
  - Hospital Maison Blanche XX Bichat, Paris
  - Hospital Sainte Anne, Paris
  - Centre Hospitalier Henri laborit, Poitiers
  - Centre Hospitalier Gillaume regnier-CHGR, Rennes
  - CHU-Saint Etienne, Saint-Etienne
  - Centre Hospitalier Alpes Isere, Saint-Égrève
  - CHITS - Hôpital Chalucet, Toulon
  - CHS St. Remy, Vesoul
- Germany (6):
  - Rheinhessen-Fachklinik Alzey, Alzey
  - Vivantes Klinikum, Berlin
  - LVR- Klinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Magdeburg, Magdeburg
  - Kbo-Isar-Ampere-Klinikum Taufkirchen, Taufkirchen
- Italy (18):
  - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Bari
  - Ospedale Versilia di Camaiore, Camaiore
  - Cura Neuropsichiatria Villa Von Siebenthal, Genzano di Roma
  - P.O. di Giulianova Dipartimento di Salute Mentale Servizio di Psichiatria di Diagnosi e Cura, Giulianova
  - Mental Health Department (MDSM) ASP di Messina, Messina
  - Ospedale Niguarda, Milan
  - Dipartimento di Salute Mentale -ASL Modena, Modena
  - Centro Salute Mentale di Pesaro, Pesaro
  - Azienda Ospedaliera "Sant' Andrea" di Roma - U.O.C. di Psichiatria, Roma
  - Fondazione PTV Policlinico Tor Vergara, Roma
  - Villa Maria Dia Hospital, Rome
  - Unit Mental Health District Nº72- ASL Salerno, Salerno
  - Unita Operativa- Salute Mentale di Salerno, Salerno
  - Centro di Salute Mentale, Saluzzo
  - Ospedale Madonna del Soccorso San Bendedetto del Tronto, San Benedetto del Tronto
  - Dipartimento di Salute Mentale- ASL Napoli, San Giorgio a Cremano
  - ASL di Teramo, Teramo
- Spain (27):
  - Hospital Punta de Europa, Algeciras, Cadiz
  - Hospital Príncipe de Asturias, Alcalá de Henares
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Sant pau, Barcelona
  - Hospital del Mar, Barcelona
  - IINA (Instituto Internacional de Neurociencias Aplicadas), Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital santa Caterina -IAS, Girona
  - Hospital Campus de la Salud, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Clínico San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hermanas Hospitalarias de Málaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Son Espases, Palma
  - Hospital Parc Taulí, Sabadell
  - Hospital Sant Joan de Déu de Sant Boi, Sant Boi de Llobregat
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Provincial de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital de Vic, Vic
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Provincial de Zamora, Zamora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Such P, Bog M, Kabra MS, Jorgensen KT, de Jong-Laird AC. A Noninterventional Cohort Study Assessing Time to All-Cause Treatment Discontinuation After Initiation of Aripiprazole Once Monthly or Daily Oral Atypical Antipsychotic Treatment in Patients With Recent-Onset Schizophrenia. Prim Care Companion CNS Disord. 2021 Sep 30;23(5):20m02886. doi: 10.4088/PCC.20m02886. PMID 34592798